CLINICAL TRIAL: NCT06300775
Title: A Comparative Evaluation of Modified Hyrax Versus Quad Helix in Treatment of Children With Posterior Cross Bite: Randomized Controlled Trial
Brief Title: Evaluation of Modified Hyrax Versus Quad Helix in Treatment of Posterior Cross Bite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sally Mohamed Mosallam, phd researcher student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123789
Record Dates: First submitted 2023-10-27; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Posterior Cross Bite

STUDY DESIGN:
Intervention Model Description: Modified Hyrax Versus Quad Helix
Masking Description: no Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Hyrax (Active Comparator): Appliance used for rapid maxillary expansion
  Interventions: Device: modified hyrax
- Quad Helix (Active Comparator): Appliance used for slow maxillary expansion
  Interventions: Device: quad helix

INTERVENTIONS:
Device: modified hyrax — Appliance used for rapid maxillary expansion
  Arms: Modified Hyrax
Device: quad helix — device use for slow maxillary expansion
  Arms: Quad Helix

SUMMARY:
This study will be performed to evaluate the treatment of posterior cross-bite with modified hyrax & Quad helix appliances and to compare which one will provide better results in relation to chewing difficulty in children with posterior cross- bite in mixed dentition

DETAILED DESCRIPTION:
This study will be performed to evaluate the treatment of posterior cross-bite with modified hyrax & Quad helix appliances and to compare which one will provide better results in relation to chewing difficulty as a primary outcome of this study and also evaluate the increase in the inter maxillary width , sleep apnea and signs & symptoms of tempro-mandibular joints disorder in children with posterior cross- bite in mixed dentition Cases will be examined within a regular interval up to one year

ELIGIBILITY:
Inclusion Criteria:

* Children with posterior cross-bite in mixed dentition stage.
* Children with normal and mild growth pattern.
* Children with completely erupted upper first molars.

Exclusion Criteria:

* Children with advanced periodontal diseases.
* Children having general diseases, syndromes.
* Children with previous orthodontic.
* Children with severe horizontal growth patterns.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Chewing difficulty | one year
  the outcome will be measured by visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo univeristry, Cairo, Egypt